CLINICAL TRIAL: NCT05541289
Title: An Intermediate Size Expanded Access Program of Whole, Inactivated SARS-CoV-2 Vaccine COVAXIN™ (BBV152) in Adults Aged 18 Years and Older
Brief Title: Expanded Access Program of Whole, Inactivated COVID-19 Vaccine COVAXIN™ (BBV152) in Adults Aged 18 Years and Older
Status: No longer available | Type: Expanded Access
Sponsor: Ocugen (Industry)
Responsible Party: Sponsor
Other Study IDs: OCU-004EA
Record Dates: First submitted 2022-09-09; First posted 2022-09-15 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
Keywords: Expanded Access; EAP; COVAXIN; BBV152
MeSH Terms: conditions — COVID-19 | interventions — BBV152 COVID-19 vaccine

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: BBV152 — Single Arm; BBV152 (COVAXIN™)
  Other Names: COVAXIN

SUMMARY:
This Expanded Access, Phase 3, open label study is intended to provide access to COVAXIN™ (BBV152) to individuals who are at risk or have predisposing conditions that can lead to complications with the current immunization options against SAR-CoV-2 Virus infection.

DETAILED DESCRIPTION:
This is an open-label single-arm single-center protocol designed to provide expanded access and evaluate the safety of COVID-19 Vaccine, COVAXIN™ (BBV152) in adults, who either decline or do not qualify for current m-RNA based Covid19 vaccines and whose locations or circumstances put them at appreciable risk of exposure to SARS-CoV-2 and development of COVID-19.

Each participant will receive a 2-dose regimen of the study vaccine (SV) as an intramuscular (IM) injection in the deltoid region of the upper arm at least 28 days apart (the first dose on Day 1 and the second dose on Day 29).

Safety assessment will include monitoring: Adverse events following immunization (AEFI)

; Adverse event of special interest (AESI) defined for COVID-19 vaccines; Serious adverse event following immunization (SAEFI) ; Medically Attended Adverse Events (MAAE); Potentially Immune Mediated Medical Conditions (PIMMC).

ELIGIBILITY:
Inclusion Criteria:

1. Does not meet Inclusion/Exclusion criteria for the ongoing COVAXIN™ (BBV152), COVID-19 vaccine clinical trial(s).
2. Either:

   Has history of myocarditis or pericarditis occurred after any dose of mRNA COVID-19 vaccine OR Has a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention, including but not limited to systemic lupus erythematosus (e.g., Guillain-Barré Syndrome, rheumatoid arthritis, polyarticular juvenile idiopathic arthritis, psoriatic arthritis, ankylosing spondylitis, multiple sclerosis, systemic lupus erythematous).

   OR Unwilling to or unable to be vaccinated with the currently available vaccines due to contraindications - possible side effects such as myocarditis, pericarditis, Guillain-Barré syndrome or thromboembolic events , treating physician discretion or any other personal preference.
3. Adults, ≥ 18 years of age at time of consent, who based on the Investigator's discretion are at high risk of SARS-CoV-2 infection, defined as adults whose locations or circumstances put them at appreciable risk of exposure to SARS-CoV-2 and development of COVID-19.
4. Understands and agrees to comply with the study procedures and provides written informed consent.
5. In relatively stable health based on site Investigator's judgment, as determined by medical history, physical examination, and the following criteria:
6. Stable health for age (defined as no new conditions per medical history, new medications in a different therapeutic class, or change in daily dose of existing prescription medications within the 45 days preceding Screening). Effective treatment (to resolution) of an acute infection (e.g., urinary tract infection, cellulitis, otitis, or bronchitis) with an antibiotic within 45 days preceding Screening will not be considered a deviation from this inclusion criterion as long as the antibiotic therapy was completed at least one week prior to Screening and no signs or symptoms of the infection have been present since the completion of treatment. Any prescription change that is due to change of health care provider or insurance company, or that is made for reasons that do not reflect a change in disease status (e.g., financial considerations), as long as within the same general class of medication, will not be considered a deviation from this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site investigator, will not be considered a deviation from this inclusion criterion.
7. Participants may be on chronic or as needed medications if, in the opinion of the Investigator, these pose no additional risk to participant safety and their use is not for management of a worsening of medical diagnosis or condition.
8. Female participants of childbearing potential may be enrolled in the study if the participant fulfills all the following criteria:

   * Have a negative pregnancy test at Baseline and prior to each study dose.
   * Have agreed to continue adequate contraception during the study and for 3 months following the second dose of the study vaccine.
   * Is not currently breastfeeding. Adequate female contraception is defined as consistent and correct use of a Food and Drug Administration (FDA) approved contraceptive method in accordance with the product label.
9. Agrees to not take part in any other COVID-19 vaccine clinical trial for the duration of the study.

Exclusion Criteria:

1. Is acutely ill or febrile 72 hours prior to or at Baseline. Fever is defined as a body temperature ≥ 38.0°C/100.4°F. Participants meeting this criterion may be rescheduled when the fever has resolved and there has not been any symptoms for > 14 days before enrollment.
2. Is pregnant or breastfeeding.
3. Known or suspected allergy or history of anaphylaxis, urticaria, or other significant adverse reaction to the vaccine or any of its components.
4. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
5. History of heparin-induced thrombocytopenia (HIT) withing 90 days prior enrollment.
6. Previous vaccination with any coronavirus vaccine within 6 months prior enrollment.
7. Has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to Baseline (for corticosteroids ≥20 milligram (mg)/day of prednisone equivalent).
8. Immunosuppressive or immunodeficient state, asplenia, recurrent severe infections (HIV-positive participants with CD4 count ≥350 cells/mm3 and an undetectable HIV viral load within the past year [low level variations from 50-500 viral copies which do not lead to changes in antiretroviral therapy [ART] are permitted]).

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Woods, Langhorne, Pennsylvania, United States

REFERENCES:
- See also: Non-Human Primate Efficacy Study Immunogenicity and protective efficacy of inactivated SARS-CoV-2 vaccine candidate, BBV152 in rhesus macaques — https://www.nature.com/articles/s41467-021-21639-w
- See also: Persistence of immunity and impact of third dose of inactivated COVID-19 vaccine against emerging variants — https://www.nature.com/articles/s41598-022-16097-3